CLINICAL TRIAL: NCT04502407
Title: IIT2019-20-Zumsteg-HPVOPC: Phase II Trial of De-Intensified Post-operative Chemoradiation Following Robotic Surgery for HPV-positive Oropharyngeal Cancer
Brief Title: Trial of De-Intensified Post-operative Chemoradiation Following Robotic Surgery for HPV-positive Oropharyngeal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Zachary Zumsteg, Assistant Professor, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2019-20-Zumsteg-HPVOPC
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: cisplatin; chemoradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- De-intensified Cisplatin-based Chemoradiation (Experimental): This is a non-randomized study, with all patients undergoing de-intensified post-operative cisplatin-based chemoradiation. Dosage level and duration of administration will be determined by whether the patient is high risk or not as assessed by the treating investigator.
  Interventions: Radiation: Cisplatin-based Radiation Therapy; Drug: Cisplatin Chemotherapy

INTERVENTIONS:
Radiation: Cisplatin-based Radiation Therapy — * High risk patients who are patients with positive margins, extranodal extension, or ≥5 positive lymph nodes will receive radiation dose of 50 Gy in 25 fractions over 5 cycles on Days 1, 8, 15, 22, and 29 of radiation treatment.
  * All other patients will receive radiation dose of 30 Gy in 15 fractions over 3 cycles on Days 1, 8 and 15 of radiation treatment.
Drug: Cisplatin Chemotherapy — * High risk patients who are patients with positive margins, extranodal extension, or ≥5 positive lymph nodes will receive 5 cycles of weekly chemotherapy of cisplatin 40mg/m2 given intravenously (IV) on Days 1, 8, 15, 22, and 29 of radiation.
  * All other patients will receive 3 cycles of weekly chemotherapy of cisplatin 40mg/m2 given intravenously (IV) on Days 1, 8 and 15 of radiation.

SUMMARY:
This study will enroll patients with HPV-associated oropharyngeal cancer, undergoing resection of all gross visible disease at the primary site and in the lymph nodes. A total of 40 patients who have had or will require surgery to remove cancer cells prior to starting chemoradiation may be enrolled. All eligible patients will receive de-intensified cisplatin-based chemoradiation, with high-risk patients receiving a higher dose and longer treatment period than other patients on the study. The study will assess whether a de-intensified version of standard chemoradiation treatment will be just as effective in treating HPV-associated oropharyngeal cancer while causing less side effects than standard dosing.

DETAILED DESCRIPTION:
This is a single arm phase II study that will enroll patients with HPV-associated oropharyngeal cancer, undergoing resection through trans-oral robotic surgery (TORS) of all gross visible disease at the primary site and in the lymph nodes. A total of 36 patients at Cedars-Sinai Medical Center and its affiliates (Tower Hematology-Oncology, Torrance Memorial Physician Network) who have had or will require surgery to remove cancer cells prior to starting chemoradiation may be enrolled. All eligible patients will receive de-intensified cisplatin-based chemoradiation, with high-risk patients receiving a higher dose and longer treatment period than other patients on the study. The treatment period will last 3 to 5 weeks depending on whether the patient is considered high-risk or not. The study will assess whether a de-intensified version of standard chemoradiation treatment will be just as effective in treating HPV-associated oropharyngeal cancer while causing less side effects than standard dosing.

ELIGIBILITY:
Inclusion Criteria:

1. AJCC 8th edition T0-3N0-2 p16-positive oropharyngeal (tonsil, base of tongue, glossotonsillar sulcus, soft palate, oropharyngeal wall) squamous cell carcinoma or squamous cell carcinoma of unknown primary involving the cervical lymph nodes. Cytologic diagnosis from a cervical lymph node is sufficient for diagnosis in the presence of clinical evidence of a primary tumor in the oropharynx.
2. For patients with pT0 tumors (unknown primary), there must be at least one metastatic lymph node present in cervical level II.
3. p16 should be strongly and diffusely positive in the nuclear and cytoplasmic component in greater than 70% of the tumor cells.
4. Have undergone or will undergo gross total resection of all known disease in the head and neck via transoral robotic surgery. For patients with unknown primary tumors, a minimum of an ipsilateral tonsillectomy and base of tongue resection is required.
5. Have undergone or will undergo neck dissection.
6. Have at least one of the following after surgery:

   * Pathologic stage T3
   * 2 or more positive lymph nodes
   * At least one lymph node >3cm
   * Lymphovascular invasion
   * Perineural invasion
   * Extranodal extension
   * Close/positive margins: Close margins are considered <3mm from the peripheral margins and <1mm from the deep margin on the en bloc specimen, unless the area of close margin is re-resected and without carcinoma.
7. Age ≥ 18 years old
8. ECOG performance status 0 or 1 within 56 days of start of chemoradiation.
9. Women of childbearing potential require a negative serum or urine pregnancy test within 28 days prior to start of chemoradiation.
10. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
11. Adequate hematologic and renal function within 30 days of start of chemoradiation, defined as:

    * Hemoglobin ≥ 9.0 g/dL
    * Platelets ≥ 100, 000 cells/mm3
    * ANC ≥ 1.5 X 109/L
    * Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
    * Aspartate aminotransferase/alanine aminotransferase ≤ 3.0 x upper limit of normal (ULN)
    * Serum creatinine ≤1.5 x upper limit of normal (ULN) OR a calculated creatinine clearance ≥60 mL/min

Exclusion Criteria:

1. AJCC 8th edition pT4 or cN3 disease.
2. Radiologic or clinical evidence of distant metastasis.
3. Recurrent disease.
4. Inability to achieve gross total resection at time of surgery.
5. Greater than 56 days (8 weeks) after surgical resection of the primary site.
6. Prior radiation to the head and neck > 30 Gy.
7. Prior active invasive (not in situ) malignancy within the prior 2 years, excluding cutaneous basal cell or squamous cell carcinoma, low or intermediate risk prostate cancer, papillary thyroid cancer, AJCC 8th edition stage I-II breast cancer, or low grade non-Hodgkin lymphoma
8. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
   * Transmural myocardial infarction within the last 6 months
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   * Hepatic insufficiency resulting in clinical jaundice and/or known coagulation defects
   * Uncontrolled Acquired Immune Deficiency Syndrome (AIDS), defined as a CD4 count < 200 at screening or an AIDS-defining opportunistic infection within the last 6 months.
9. Moderate to severe hearing loss.
10. Active connective tissue disease (e.g. systemic lupus erythematous, scleroderma) requiring immunosuppression.
11. Pregnant or breast-feeding women.
12. Prior allergic reaction to cisplatin.
13. Live vaccines within 30 days prior to the first dose of chemoradiation. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral vaccine). Season influenza vaccines for injection are generally killed virus vaccines and are allowed; however intranasal influenza vaccines (e.g. Flu-Mist®) are live attenuated vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
2-Year Progression-Free Survival (PFS) | 2 years
  Proportion of patients alive and without evidence of local, regional, or distant recurrence at 2 years from study enrollment.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  Proportion of patients alive, based on time from enrollment to death from any cause.
Local Control | 2 years
  Proportion of patients without recurrence at the primary site, based on time from enrollment to local recurrence, irrespective of prior regional or distant recurrence. Death from causes unrelated to cancer is a competing event.
Regional Control | 2 years
  Proportion of patients without recurrence in the cervical lymph nodes, based on time from enrollment to regional recurrence, irrespective of prior local or distant recurrence. Death from causes unrelated to cancer is a competing event.
Locoregional Control | 2 years
  Proportion of patients without local recurrence or regional recurrence, as defined above, based on the time from enrollment to the first evidence of either local or regional recurrence, irrespective of prior distant recurrence. Death from causes unrelated to cancer is a competing event.
Distant Control | 2 years
  Proportion of patients without distant recurrence, based on time from enrollment to distant recurrence, irrespective of prior local or regional recurrence. Distant metastasis includes any recurrent disease outside of the head and neck, cervical lymph nodes, or retropharyngeal lymph nodes. Death from causes unrelated to cancer is a competing event.
Cause-specific Survival | 2 years
  Proportion of patients without oropharyngeal cancer-related or treatment-related death, based on time from enrollment to death from oropharyngeal cancer or treatment. Death from other causes is a competing event.
Mean change in patient-reported outcomes using Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | 2 years
  PRO-CTCAE responses are scored from 0 to 4 (or 0/1 for absent/present), with lower scoring indicating an absence of symptoms to higher scoring reflecting higher severity of symptoms.
Mean change in patient-reported outcomes using Hearing Handicap Inventory for Adults (HHIA-S) | 2 years
  The scale ranges from 0 to 4 (0 - no, 2 - sometimes, 4- yes) for each question identifying problems with hearing loss, as self-reported by patients. The total number of points for the 25 questions range from 0 to 100, with 0 indicating no handicap to 100 indicating total handicap.
Mean change in patient-reported outcomes using European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) | 2 years
  The EORTC QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL, and six single items. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems. Most questions are scored 1 to 4, with exception to global health questions scored from 1 to 7. The raw scores are then standardized by a linear transformation, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Mean change in patient-reported outcomes using University of Michigan Xerostomia-Related Quality of Life Scale (XeQoLS) | 2 years
  XeQOLS is a patient-reported, 15-item scale that measures four domains: physical functioning, pain/discomfort, personal/psychologic functioning, and social functioning. Patient responses to all four domains are averaged, and the total scores range from 0 to 4; an increased xerostomia burden is indicated by a higher score.
Mean change in patient-reported outcomes using 5-level version of the EuroQol five dimensional instrument EQ-5D-5L | 2 years
  The EQ-5D-5L descriptive system comprises of five dimensions: (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION), with each dimension having five response levels: no problems, slight problems, moderate problems, severe problems, unable to /extreme problems - severity level of each dimension are coded from 1 to 5, respectively. The visual analog scale (EQ VAS) attached to this questionnaire records the respondent's overall self-rated perception of current health status on a vertical visual analogue scale, where the endpoints are scored from 0 to 100, 100 being the 'The best health you can imagine' and 0 indicating 'The worst health you can imagine'
Mean change in patient-reported outcomes using the MD Anderson Dysphagia Inventory (MDADI) | 2 years
  The MDADI is a patient-reported, 20-item scale that quantifies four domains: an individual's global (G), physical (P), emotional (E), and functional (F) perceptions of their swallowing ability. Two summary scores can be obtained from the MDADI: 1) global and 2) composite. The global scale is a single question, scored individually, to assess the overall impact that swallowing abilities have on quality of life ("my swallowing impacts my day-to-day life"). The composite MDADI score summarizes overall performance on remaining 19-items of the MDADI, as a weighted average of the physical, emotional, and functional subscale questions. Summary and subscale MDADI scores are normalized to range from 20 (extremely low functioning) to 100 (high functioning). Five possible responses to the items on the MDADI are: strongly agree, agree, no opinion, disagree, and strongly disagree, and scored on a scale of 1 to 5 respectively.
Progression-free survival (PFS) in high-risk and intermediate risk patient subgroups | 2 years
  The difference between the proportion of patients alive and without evidence of local, regional, or distant recurrence at 2 years from study enrollment, in high-risk and intermediate subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary S Zumsteg, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (4):
- United States (4):
  - Tower Hematology-Oncology, Beverly Hills, California
  - Cedars-Sinai Medical Center (Beverly - Main Site), Los Angeles, California
  - Valley Oncology Medical Group, Tarzana, California
  - Torrance Memorial Physician Network Cancer Care, Torrance, California